CLINICAL TRIAL: NCT04525781
Title: Clinicoepidimiological Study and Clinical Outcome in Patients With Urinary Bladder Cancer at Assuit University Hospital From 2015 to 2019(Hospital Based Study)
Brief Title: Clinicoepidimiological Study and Clinical Outcome in Patients With Urinary Bladder Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rehab Osama Abdelmaboud, Principal Investigator, Assiut University
Other Study IDs: Urinary bladder cancer.
Record Dates: First submitted 2020-08-20; First posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Urinary Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
To pinpoint the clinical ,epidimiological factors and clinical outcomes in urinary bladder cancer patients attending to our department during 5 years period between 2015-2019.

DETAILED DESCRIPTION:
Bladder cancer is the ninth most common cancer throughout the world. The incidence of bladder cancer is three to four times greater in men than in women. However, women are diagnosed with more advanced disease at presentation and have less favorable outcomes after treatment. Statistical data show that between 2002 and 2012, worldwide, the number of bladder cancers increased from 375.000 to about 430.000 , while the mortality increased from 145.000 patients in 2002 up to 165.000 patients in 2012. In the United States, bladder cancer is the fourth most common cancer in males with an age-adjusted incidence rate of 37.3/100,000 person years (PY) using the US standard population.

In developed countries, over 90% of the bladder cancer cases diagnosed are transitional cell carcinoma (TCC), with squamous cell carcinoma (SCC), adenocarcinomas, and rare types of bladder cancer comprising the remaining 10% of bladder cancer cases.

Exposures to tobacco smoke, occupational toxins, and environmental sources of heavy metals such as arsenic are the major reported risk factors for TCC.

Unlike TCC, the main risk factors for SCC are not environmental exposures, but exposure to infectious agents. Age, smoking, tumor stage and the treatment modalities such as surgery and adjuvant chemotherapy were proved to affect the overall survival in patients with urinary bladder cancer. Our study may give an important evidence about clinical, epidemiological factors and clinical outcomes in urinary bladder cancer patients at Assuit University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* age 18 :70
* Histologically proved urinary bladder carcinoma

Exclusion Criteria:

* Age less than 18 or more than 70
* Patient not documented having bladder carcinoma with biopsy [cysyoscopic or operative]
* Patient with synchronous or metachronous double primary

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: study initialy including about 150 patients with urinary bladder cancer.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
comparison of response in non muscle invasive,muscle invasive and metastatic bladder cancer. | baseline
  Analysis of patients data including risk factors and treatment and detection of response in each stage.

SECONDARY OUTCOMES:
Survival in bladder cancer in different stages | baseline

REFERENCES:
- [Background] Parkin DM, Bray F, Ferlay J, Pisani P. Global cancer statistics, 2002. CA Cancer J Clin. 2005 Mar-Apr;55(2):74-108. doi: 10.3322/canjclin.55.2.74. PMID 15761078
- [Background] Dobruch J, Daneshmand S, Fisch M, Lotan Y, Noon AP, Resnick MJ, Shariat SF, Zlotta AR, Boorjian SA. Gender and Bladder Cancer: A Collaborative Review of Etiology, Biology, and Outcomes. Eur Urol. 2016 Feb;69(2):300-10. doi: 10.1016/j.eururo.2015.08.037. Epub 2015 Sep 4. PMID 26346676
- [Background] Murta-Nascimento C, Schmitz-Drager BJ, Zeegers MP, Steineck G, Kogevinas M, Real FX, Malats N. Epidemiology of urinary bladder cancer: from tumor development to patient's death. World J Urol. 2007 Jun;25(3):285-95. doi: 10.1007/s00345-007-0168-5. PMID 17530260
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] Malats N, Real FX. Epidemiology of bladder cancer. Hematol Oncol Clin North Am. 2015 Apr;29(2):177-89, vii. doi: 10.1016/j.hoc.2014.10.001. PMID 25836927
- [Background] Zhao M, He XL, Teng XD. Understanding the molecular pathogenesis and prognostics of bladder cancer: an overview. Chin J Cancer Res. 2016 Feb;28(1):92-8. doi: 10.3978/j.issn.1000-9604.2016.02.05. PMID 27041931
- [Background] Jemal A, Murray T, Ward E, Samuels A, Tiwari RC, Ghafoor A, Feuer EJ, Thun MJ. Cancer statistics, 2005. CA Cancer J Clin. 2005 Jan-Feb;55(1):10-30. doi: 10.3322/canjclin.55.1.10. PMID 15661684
- [Background] Lynch CF, Cohen MB. Urinary system. Cancer. 1995 Jan 1;75(1 Suppl):316-29. doi: 10.1002/1097-0142(19950101)75:1+3.0.co;2-t. PMID 8001003
- [Background] Golka K, Wiese A, Assennato G, Bolt HM. Occupational exposure and urological cancer. World J Urol. 2004 Feb;21(6):382-91. doi: 10.1007/s00345-003-0377-5. Epub 2003 Nov 26. PMID 14648102
- [Background] Chen CJ, Chuang YC, You SL, Lin TM, Wu HY. A retrospective study on malignant neoplasms of bladder, lung and liver in blackfoot disease endemic area in Taiwan. Br J Cancer. 1986 Mar;53(3):399-405. doi: 10.1038/bjc.1986.65. PMID 3964542
- [Background] Shokeir AA. Squamous cell carcinoma of the bladder: pathology, diagnosis and treatment. BJU Int. 2004 Jan;93(2):216-20. doi: 10.1111/j.1464-410x.2004.04588.x. PMID 14690486
- See also: Surveillance Epidemiology End Results. Cancer Stat Facts Sheet — http://seer.cancer.gov/statfacts/.